CLINICAL TRIAL: NCT06311331
Title: Prospective Evaluation of Clinical and Radiographic Outcomes Following Total Talus Replacement (PROCLAIM): A Multicenter, Single Arm, Prospective, Post-approval Study for Patients Who Received the restor3d TTR Device to Evaluate Safety and Probable Benefit
Brief Title: Prospective Evaluation of Clinical and Radiographic Outcomes Following Total Talus Replacement (PROCLAIM)
Status: Enrolling by invitation | Type: Observational
Sponsor: Restor3D (Industry)
Collaborators: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: restor3d-007
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Avascular Necrosis of the Talus; Talar Osteochondral Defect of Ankle; Talar Dysfunction
Keywords: Avascular necrosis; Talus; Ankle joint
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Total Talus Replacement: 50 subjects receiving the Total Talus Replacement device
  Interventions: Device: Total Talus Replacement (TTR)

INTERVENTIONS:
Device: Total Talus Replacement (TTR) — The restor3d patient-specific TTR Implant and Instrumentation System is designed to replace a native talus bone that has been affected by a disease state or injury. The implant is an additively manufactured Cobalt Chromium alloy (ASTM F3213) construct produced by laser powder bed fusion. The data-driven design of the implant enables the patient to salvage their joint while maintaining ankle range of motion, reducing pain and improving physical function.

SUMMARY:
This is a Humanitarian Device Exemption (HDE) approved device. The purpose of this study is to evaluate the continued safety and probable benefit of the restor3d Total Talus Replacement device in commercial use.

ELIGIBILITY:
Inclusion Criteria:

* ≥22 Years of Age
* Scheduled to receive TTR implant for one of the following indications:
* Avascular necrosis of the talus
* Avascular necrosis of the talus in addition to talar collapse, cysts or non-union
* Large, uncontained, unstable, or cystic talar osteochondral defects with risk of collapse or talar osteochondral defects not responsive to traditional treatments
* Nonunion following talar fracture or talar extrusion, unresponsive to more conservative treatments
* Have not had a prior Total Talus Replacement device implanted
* Not planning to receive bilateral Total Talus Replacement devices
* Subject signs a written informed consent form (ICF) prior to the surgical procedure

Exclusion Criteria:

* Surgical procedures other than those listed in the indications for use.
* Use of implant greater than 6 months from date of patient's preoperative CT scan.
* Degenerative changes in the tibiotalar, subtalar or talonavicular joints.
* Gross deformity in sagittal or coronal planes. More than 15 degrees of varus or valgus deformity in the coronal plane, or more than 50% subluxation anteriorly or posteriorly of the talus in the sagittal plane
* Patients with an active local or systemic infection.
* Osteonecrosis of the calcaneus, distal tibia or navicular.
* Known history of existing malignancy, or any systemic infection, local infection, or skin compromise at the surgical site.
* Blood supply limitations and previous infections that may prevent healing.
* Physical conditions that would eliminate adequate implant support or prevent healing, including inadequate soft tissue coverage.
* Conditions which may limit the patient's ability or willingness to restrict activities or follow directions postoperatively during the healing period.
* Presence of neurological deficit which would prevent patient postoperative compliance.
* Patients with foreign body sensitivity, suspected or documented material allergy or intolerance. Where material sensitivity is suspected, appropriate tests should be conducted, and sensitivity ruled out prior to implantation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥22 years of age) who will receive a restor3d Total Talus Replacement device under an approved HDE for one of the indications listed on the Instructions for Use (IFU) and who do not have a contraindication (see Inclusion and Exclusion Criteria)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who pass a composite of safety and probable benefit outcomes | At 5 years compared to baseline
  The primary endpoint for this post approval study is a composite of safety and probable benefit.
  The safety endpoint is defined by the absence of device-related SAE and subsequent secondary surgical intervention (SSSI) on the affected joints.
  The probable benefit endpoint is defined as joint salvage with the restor3d device still in place.
  This composite endpoint will be evaluated by determining the proportion of patients who do not have a device-related SAE or SSSI, AND have the restor3d implant in place at 5 years.

SECONDARY OUTCOMES:
Change in perceived pain from baseline | At 5 years compared to baseline
  Scores on the 11-point Pain Numeric Rating Scale (NRS) rated from 0-10 where higher scores indicate worse pain
Change in Foot and Ankle Outcome Score (FAOS) Composite score from baseline | At 5 years compared to baseline
  Foot and Ankle Outcome Score (FAOS) is a 42-item questionnaire with 5 subscales: pain (9 items), other symptoms (7 items), activities of daily living (ADL) (17 items), sports/recreation (5 items), and quality of life (4 items). Each question is graded from 0 to 4 on a 5-point Likert scale (none, mild, moderate, severe, and extreme problems). Composite FAOS scores include all 42-items across the 5 subscales, scored together to provide one comprehensive value. The FAOS composite score ranges from 0 to 100 where a score of 0 indicates the worst possible symptoms, and a score of 100 indicates no symptoms.
Change in Foot and Ankle Outcome Score (FAOS) pain subscale score from baseline | At 5 years compared to baseline
Change in Foot and Ankle Outcome Score (FAOS) other symptoms subscale score from baseline | At 5 years compared to baseline
Change in Foot and Ankle Outcome Score (FAOS) activities of daily living (ADL) subscale score from baseline | At 5 years compared to baseline
Change in Foot and Ankle Outcome Score (FAOS) sports/recreation subscale score from baseline | At 5 years compared to baseline
Change in Foot and Ankle Outcome Score (FAOS) quality of life (QOL) subscale score from baseline | At 5 years compared to baseline
Change in ankle range of motion (ROM) from baseline | At 5 years compared to baseline
  Ankle ROM will be evaluated using a goniometer to determine the change in degrees of plantarflexion and dorsiflexion
Proportion of procedure-related Serious Adverse Events | At 5 years compared to baseline
  Procedure-related Serious Adverse Event will be defined as the number of patients who have a procedure-related event including: death, life-threatening condition, hospital admission (initial or prolonged), disability or permanent damage, or required intervention to prevent permanent impairment or damage.
Proportion of Adverse Events | At 5 years compared to baseline
  Adverse Event will be defined as the number of patients who have a non-serious, unexpected procedure- or device-related event before 5 years post-implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina Research Institute, Inc., Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided